CLINICAL TRIAL: NCT04080505
Title: Does the Use of Pre-operative SSKI Actually Reduce Vascularity and Improve Surgical Outcomes for Total Thyroidectomy in Graves' Disease?
Brief Title: Does Potassium Iodide (SSKI) Reduce Vascularity in Graves' Thyroidectomy?
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Jennifer Kuo, Assistant Professor of Surgery, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAO3312
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Graves Disease
MeSH Terms: conditions — Graves Disease | interventions — Potassium Iodide

STUDY DESIGN:
Intervention Model Description: All participants complete a baseline neck ultrasound no less than 7 days prior to surgery, to obtain vascular flow imaging. Participants are then randomized to receive 7 days of pre-operative SSKI or not receive any drug. In the practice at Columbia, all patients with Graves' disease receive SSKI preoperatively, though this is not standard practice across the country, thus the 'no drug' group is experimental for research.
  All participants complete a second ultrasound on the operating table before surgery, to assess for change in vascularity (experimental, as not all patients receive intra-operative ultrasounds before surgery). Both ultrasounds are performed by the surgeon.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SSKI (Potassium Iodide) (Active Comparator): Participants randomized to receive 7 days of pre-operative SSKI
  Interventions: Drug: SSKI- Potassium Iodide
- NO SSKI (No Intervention): Participants randomized to not receive any drug pre-operative

INTERVENTIONS:
Drug: SSKI- Potassium Iodide — 1g/mL, 2 drops orally 3 times a day for 7 days before surgery
  Arms: SSKI (Potassium Iodide)

SUMMARY:
The purpose of this research is to find out if SSKI (Potassium Iodide) reduces vascularity (the number and concentration of blood vessels) and improves how well patients do after surgery for removal of their whole thyroid gland in Graves' disease (an autoimmune disease that is a common cause of hyperthyroidism).

DETAILED DESCRIPTION:
Patients with Graves' disease and goiters tend to have very vascular thyroid glands, which increases operative bleeding risks/rates. Many surgeons treat these patients with preoperative SSKI which is believed to decrease the vascularity, which in turn may decrease bleeding risks. However, there has been no quantitative data published on whether this is a real effect with true clinical benefit, in either animal or human models with SSKI. There have been some studies in Europe studying Lugol's solution, a different formulation of iodine, which show some decreased vascularity using color Doppler or measurements of CD34 cells.

ELIGIBILITY:
Inclusion Criteria:

* individuals diagnosed with Graves' disease undergoing total thyroidectomy for cure of disease.

Exclusion Criteria:

* no Graves' disease
* < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-02-10 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Kuo, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants withdrew from the study prior to randomization.
Period: Overall Study
Arm/Group | SSKI (Potassium Iodide) | No SSKI
Started | 16 | 11
Completed | 16 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SSKI (Potassium Iodide) | NO SSKI | Total
Number analyzed (Participants) | 16 | 11 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 9 | 23
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 8 | 3 | 11
  Black or African American | 2 | 2 | 4
  Asian | 0 | 0 | 0
  Hispanic or Latino | 0 | 1 | 1
  Other | 0 | 0 | 0
  Not reported | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 16 | 11 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change in Vascular Flow From Baseline
Description: Using 3D imaging software, the investigators will quantify the vascular flow in the ultrasound images and compare baseline images with the operating room (OR) images to assess if there is a difference in vascular flow between those timepoints. Vascular flow will be quantified using percent (%) surface area. This calculation will be done by a computer algorithm.
Time Frame: From Baseline to Immediately Before Surgery
Population: Data was not collected and therefore cannot be analyzed.
Arm/Group | SSKI (Potassium Iodide) | No SSKI
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | SSKI (Potassium Iodide) | No SSKI
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/11
Other Adverse Events (participants affected / at risk) | 0/16 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT04080505/Prot_SAP_000.pdf